CLINICAL TRIAL: NCT05822323
Title: Retrospective Evaluation Of The Effect Of Botulinum Toxin-A Injection Applied To The Mental Muscle On Free Gingival Graft Operation: A Randomized Controlled Clinical Study
Brief Title: Effect of Botulinum Toxin-A on Free Gingival Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kevser Sokmen (Other)
Responsible Party: Sponsor-Investigator, Kevser Sokmen, Asisstant Professor, Alanya Alaaddin Keykubat University
Organization: Alanya Alaaddin Keykubat University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AlanyaAKÜ
Record Dates: First submitted 2023-04-06; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Gingival Recession, Localized
Keywords: Gingival recession; free gingival graft; mental muscle; Botulinum Toxin-A; keratinized gingiva
MeSH Terms: conditions — Gingival Recession | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: The study was carried out on 40 lower incisors of 40 patients who applied to the Fırat University Faculty of Dentistry Department of Periodontology between the years of 2019 and 2021, who had Miller class III gingival recession in their lower 1st incisors, and were treated with FGG operation due to insufficient amount of keratinized gingiva. The patients were divided into 2 groups as randomized controlled.
  Control group (FGG) (n:20): The patients in this group only underwent the FGG operation.
  Study group (FGG+BTX) (n:20): The patients in this group received 5 U BTX-A injection into the mental muscle immediately after the FGG operation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (FGG) (Experimental): The patients in this group only underwent the FGG operation.
  Interventions: Procedure: free gingival graft
- Study group (FGG+BTX) (Active Comparator): The patients in this group received 5 U BTX-A injection into the mental muscle immediately after the FGG operation.
  Interventions: Other: BTX-A; Procedure: free gingival graft

INTERVENTIONS:
Other: BTX-A — Vials of 100 U Allergan Botox® (Allergan, Inc., Irvine, California) were diluted with 2 ml of physiological saline and made ready for use. The midline was determined at the mentum region. 5 U of BTX-A was injected into the mental muscle approximately 1 cm away from the chin tip and the midline
  Other Names: 100 U Allergan Botox®; Allergan, Inc., Irvine, California; Botox
  Arms: Study group (FGG+BTX)
Procedure: free gingival graft — The mandibular first incisor was treated with FGG operation due to Miller class III gingival recession and insufficient amount of keratinized gingiva.

SUMMARY:
The aim of this study was to examine the effects of Botulinum Toxin-A (BTX-A) injection to the mental muscle on the free gingival graft (FGG) operation. Forty patients with Miller class III gingival recession and keratinized gingival insufficiency in their lower 1st incisors were divided into 2 groups as FGG operation (n=20) and 5 unit (U) BTX-A injection into the mental muscle immediately after FGG operation (n=20). Periodontal parameters (plaque index (PI), gingival index (GI), probing pocket depth (PPD), keratinized gingival amount (KGA), attached gingival amount (AGA)) were measured from the lower 1st incisors at the beginning and at the 1st, 3rd and 6th months after the operation, clinical attachment level (CAL), gingival thickness (GT), gingival recession amount (GRA), gingival recession width (GRW) and root closure percentage (RCP (%)) were evaluated. There was no statistically significant difference in terms of PI and GI levels (p>0.05). The PPD levels of the study group at the postoperative 3rd month was found to be statistically significantly lower than the control group (p<0.05). While the change in GT and RCP (%) levels were found to be statistically significantly higher than the control group, the change in GRW and CAL levels were statistically significantly lower (p<0.05). According to the results of this study, it can be stated that BTX-A injection applied to the mental muscle after FGG operation may have positive effects in terms of KGA, AGA, GT, RCP (%), GRW and CAL parameters.

DETAILED DESCRIPTION:
INTRODUCTION The FGG operation is a versatile surgical procedure that is frequently used in the treatment of gingival recessions to increase the width of the attached gingiva, the depth of the vestibule and to close the open root surface. While it is a more successful method in closing the open root surface in patients with Miller class I and II gingival recessions without bone loss, the same success cannot be observed in patients with Miller class III and IV gingival recessions with bone loss in the interdental area. The most important factors affecting the success of the FGG operation are the ensurement of the nourishment of the graft by maintaining the blood supply and the ensurement of graft immobility in the early recovery period by blocking the return of the dissected muscle attachments to their original position. Insufficient blood supply to the recipient bed where the graft is placed causes necrosis in the graft. In this case, there is a risk that the root surface cannot be completely covered. In addition, due to the desire of the dissected muscle attachments to return to their original position, there is a risk of not being able to achieve the desired amount of keratinized band increase.

Botox (BTX) is a toxin obtained from the Clostridium Botulinum bacteria and is a microbial protein that shows its effect by blocking neuromuscular activity. Immunologically, there are 8 different serotypes of BTX (A, B, C1, C2, D, E, F, G). Serotype A is the most potent serotype and the first form used in medicine. BTX-A is an agent used in medicine and dentistry for therapeutic purposes as well as cosmetic purposes. In the field of dentistry, it is preferred as a treatment method in many pathological conditions such as oromandibular dystonia, bruxism, asymmetry due to facial paralysis, temporomandibular joint (TMJ) disorders, gummy smile, and orange peel-looking jaw. There are studies showing that BTX application causes vasodilation in the blood vessels of the injected area; increasing the amount of blood flow and oxygen delivery at the vascular, tissue, cell and molecular levels in the region. It has been reported that this effect eliminates the risk of the necrosis of the graft whose blood connection was cut due to the increased blood supply in the region and also contributes to flap viability.

The mental muscle is a pair of muscles on the right and left, starting from the jawbone at the apical level of the incisors, moving downwards, and ending at the skin. The contraction of the mental muscle, which provides the vertical support of the lower lip; raises the lower lip and chin, creating a sullen and sad expression on the face. Due to the mental muscle ending at the skin, excessive activity of the muscle causes an indented appearance of the chin, which is called the orange peel. BTX injection applied to the mental muscle contributes to the improvement of the orange peel appearance by reducing the excessive activity of the muscle.

The aim of this retrospective study was to evaluate the effects of BTX-A injection to the mental muscle on patients with Miller class III gingival recession in their lower 1st incisors who underwent the FGG operation due to insufficient keratinized gingiva, on the basis of clinical periodontal parameters. Due to the fact that BTX-A injection applied to the mental muscle increases the blood supply of the region and decreases mental muscle activity suggests that it will positively affect the clinical periodontal parameters.

MATERIAL AND METHODS This study, which was approved by the Ethics Committee of Fırat University Medical Faculty Clinical Research Ethics Committee with the number 12/27 on 01.08.2019, was supported by the Fırat University Scientific Research Projects Management Unit with the project number DHF.19.10.

Study Population The study was carried out on 40 lower incisors of 40 patients who applied to the Fırat University Faculty of Dentistry Department of Periodontology between the years of 2019 and 2021, who had Miller class III gingival recession in their lower 1st incisors, and were treated with FGG operation due to insufficient amount of keratinized gingiva. The patients were divided into 2 groups as randomized controlled.

Control group (FGG) (n:20): The patients in this group only underwent the FGG operation.

Study group (FGG+BTX) (n:20): The patients in this group received 5 U BTX-A injection into the mental muscle immediately after the FGG operation.

Study Design In order to maintain the standardization of the study; it was made sure that the FGG operation, which is one of the treatment methods for gingival recession, and the BTX-A injection applied to the mental muscle were performed by the same physician (KS). In order to eliminate biased behavior, an experienced physician (TTY) who did not know which group the patients belonged to performed all clinical periodontal measurements. The study was terminated after the retrospective evaluation of the clinical periodontal parameters recorded in the patient follow-up forms at the baseline, 1st, 3rd and 6th month of the study period.

Clinical Procedure Non-Surgical Periodontal Treatment In this retrospective evaluation study; patients included were applied phase I periodontal treatment (detertrage and subgingival curettage), which is routinely applied in the clinic, before each surgical procedure and were also given oral hygiene training. The study protocol was explained to patients undergoing the FGG operation and FGG+BTX application and written informed consent was obtained from each individual prior to clinical periodontal examination.

Clinical Measurements PI, GI, PPD, KGA, AGA, CAL, GRA, GRW levels were measured at the baseline and at the postoperative 1st, 3rd and 6th month; GT parameters were measured at the baseline and the postoperative 6th month with a William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA) with a 0.5 mm diameter. The RCP (%) was calculated using the formula below at the postoperative 6th month.

Baseline GRA - Postoperative 6th month GRA RCP (%) = --------------------- X 100 Baseline GRA

In order to provide standardization, clinical measurements of the study area were obtained from the reference point chosen as the midbuccal surface. In cases where the FGG operation was performed on both lower first incisors, one of the teeth were chosen at the baseline and measurements were made from the same tooth throughout the study period.

Surgical Procedure The surgical procedure was started by applying infiltrative local anesthesia (2% lidocaine, 1/100.000 epinephrine) to the operation area. The initial horizontal incision was made on the Mucogingival line with a number 15 scalpel. This incision was deepened in the apical direction with sharp dissections. The recipient bed size was prepared in accordance with the graft size which was determined as 7 mm in the apico-coronal direction and with a distance of 3 mm from the graft edges in all directions. Deepitelization of the gingiva remaining in the coronal part and root surface straightening of the lower incisors were performed. The recipient bed preparation was completed by washing the operation area with 0.9% sterile saline. The graft area was determined as the palatal region, which does not contain rugae, between the mesial of the first molar and the distal of the canine in the upper jaw. After local infiltrative anesthesia (2% lidocaine, 1/100.000 epinephrine) application to the palate region, the graft was obtained with a number 15 scalpel. Bleeding in the palate area was controlled by applying pressure with moist gauze for 5 minutes. The excess fat tissue on the inner surface of the graft was cleaned on a moist sponge with a sharp scalpel or curved-tipped tissue scissors and the fixation phase was started at the recipient site. The graft was fixed to the recipient bed with the minimum number of monofilament non-resorbable 5-0 polypropylene (Katsan, İzmir, Turkey) sutures at the most coronal region of the crestal bone. Vials of 100 U Allergan Botox® (Allergan, Inc., Irvine, California) were diluted with 2 ml of physiological saline and made ready for use. The midline was determined at the mentum region. 5 U of BTX-A was injected into the mental muscle approximately 1 cm away from the chin tip and the midline. Amoxicillin + clavulanic acid 1000 mg (2 times a day), dexketoprofen 25 mg (2 times a day) and 0.12% chlorhexidine gluconate mouthwash (3 times a day) were prescribed to each patient to control the risk of post-operative pain and infection. It was recommended that the patients brush the areas other than the operation site 2 times a day, 1 day after the operation. It was recommended to gently clean the graft surface with the help of a cotton swab soaked in mouthwash. The sutures were removed on the post-operative 21st day. Photographs of the recipient area were recorded at the baseline and the postoperative 1st, 3rd, and 6th month of each patient included in the study.

Statistical Reviews While evaluating the recorded findings in this retrospective study, the IBM SPSS Statistics 22 program was used for statistical analysis. The suitability of the parameters to the normal distribution was evaluated with Kolmogorov-Smirnov and Shapiro Wilks tests and was determined that the parameters did not show normal distribution. The Mann Whitney U test was used for the comparison of the parameters between the two groups, and the Friedman test (post hoc Wilcoxon sign test) was used for comparisons within each group. Spearman's rho correlation analysis was used to evaluate the correlations between the parameters. Significance was evaluated at the p<0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* systemically healthy
* Not having the habit of using drugs that may adversely affect wound healing
* Non-mobile teeth
* No previous surgical intervention in the operation area
* No smoking habit.

Exclusion Criteria:

* Pregnant women and
* Women in the lactation period
* Mobile teeth

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Plaque İndex | baseline plaque index
  According to the plaque index (Silness& Löe, 1964); 0: There is no plaque on the gingival margin when visualized and examined with a probe.
  1. There is plaque in the form of a film attached to the free gingival margin and adjacent tooth surface, which cannot be noticed with the naked eye, but can be seen with the help of a probe.
  2. There is moderate plaque in the gingival pocket and on the tooth surface adjacent to the gingival margin, which can be seen with the naked eye.
  3. There is dense plaque on the gingival pocket and the tooth surface adjacent to the gingival margin, the interdental area is completely filled with plaque.
Plaque İndex | Change from plak index at 1 months
  According to the plaque index (Silness& Löe, 1964); 0: There is no plaque on the gingival margin when visualized and examined with a probe.
  1. There is plaque in the form of a film attached to the free gingival margin and adjacent tooth surface, which cannot be noticed with the naked eye, but can be seen with the help of a probe.
  2. There is moderate plaque in the gingival pocket and on the tooth surface adjacent to the gingival margin, which can be seen with the naked eye.
  3. There is dense plaque on the gingival pocket and the tooth surface adjacent to the gingival margin, the interdental area is completely filled with plaque.
Plaque İndex | Change from plak index at 3 months
  According to the plaque index (Silness& Löe, 1964); 0: There is no plaque on the gingival margin when visualized and examined with a probe.
  1. There is plaque in the form of a film attached to the free gingival margin and adjacent tooth surface, which cannot be noticed with the naked eye, but can be seen with the help of a probe.
  2. There is moderate plaque in the gingival pocket and on the tooth surface adjacent to the gingival margin, which can be seen with the naked eye.
  3. There is dense plaque on the gingival pocket and the tooth surface adjacent to the gingival margin, the interdental area is completely filled with plaque.
Plaque İndex | Change from plak index at 6 months
  According to the plaque index (Silness& Löe, 1964); 0: There is no plaque on the gingival margin when visualized and examined with a probe.
  1. There is plaque in the form of a film attached to the free gingival margin and adjacent tooth surface, which cannot be noticed with the naked eye, but can be seen with the help of a probe.
  2. There is moderate plaque in the gingival pocket and on the tooth surface adjacent to the gingival margin, which can be seen with the naked eye.
  3. There is dense plaque on the gingival pocket and the tooth surface adjacent to the gingival margin, the interdental area is completely filled with plaque.
Gingival index | baseline gingival index
  According to the gingival index (Löe&Silness, 1963):
  0: Healthy gingiva
  1. There is mild inflammation of the gingiva, slight discoloration and edema, but no bleeding on probing.
  2. Moderate inflammation is observed, the gingiva is red, edematous and it is shiny, there is bleeding on probing.
  3. Severe inflammation, significant redness and edema are present, ulceration may be observed, a tendency to spontaneous bleeding may be observed.
Gingival index | Change from gingival index at 1 month
  According to the gingival index (Löe&Silness, 1963):
  0: Healthy gingiva
  1. There is mild inflammation of the gingiva, slight discoloration and edema, but no bleeding on probing.
  2. Moderate inflammation is observed, the gingiva is red, edematous and it is shiny, there is bleeding on probing.
  3. Severe inflammation, significant redness and edema are present, ulceration may be observed, a tendency to spontaneous bleeding may be observed.
Gingival index | Change from gingival index at 3 months
  According to the gingival index (Löe&Silness, 1963):
  0: Healthy gingiva
  1. There is mild inflammation of the gingiva, slight discoloration and edema, but no bleeding on probing.
  2. Moderate inflammation is observed, the gingiva is red, edematous and it is shiny, there is bleeding on probing.
  3. Severe inflammation, significant redness and edema are present, ulceration may be observed, a tendency to spontaneous bleeding may be observed.
Gingival index | Change from gingival index at 6 months
  According to the gingival index (Löe&Silness, 1963):
  0: Healthy gingiva
  1. There is mild inflammation of the gingiva, slight discoloration and edema, but no bleeding on probing.
  2. Moderate inflammation is observed, the gingiva is red, edematous and it is shiny, there is bleeding on probing.
  3. Severe inflammation, significant redness and edema are present, ulceration may be observed, a tendency to spontaneous bleeding may be observed.
Probing Pocket Depth | baseline Probing Pocket Depth
  With a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA), the probe was inserted until a slight resistance was felt at the base of the pocket/sulcus, and the distance from the base of the pocket/sulcus to the free gingival margin was measured in millimeters.
Probing Pocket Depth | Change from Probing Pocket Depth at 1 month
  With a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA), the probe was inserted until a slight resistance was felt at the base of the pocket/sulcus, and the distance from the base of the pocket/sulcus to the free gingival margin was measured in millimeters.
Probing Pocket Depth | Change from Probing Pocket Depth at 3 months
  With a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA), the probe was inserted until a slight resistance was felt at the base of the pocket/sulcus, and the distance from the base of the pocket/sulcus to the free gingival margin was measured in millimeters.
Probing Pocket Depth | Change from Probing Pocket Depth at 6 months
  With a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA), the probe was inserted until a slight resistance was felt at the base of the pocket/sulcus, and the distance from the base of the pocket/sulcus to the free gingival margin was measured in millimeters.
Keratinized Gingival Amount | baseline Keratinized Gingival Amount
  The distance from the free gingival margin to the mucogingival junction was measured in millimeters with a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA).
Keratinized Gingival Amount | Change from keratinized gingival amount at 1 months
  The distance from the free gingival margin to the mucogingival junction was measured in millimeters with a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA).
Keratinized Gingival Amount | Change from keratinized gingival amount at 3 months
  The distance from the free gingival margin to the mucogingival junction was measured in millimeters with a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA).
Keratinized Gingival Amount | Change from keratinized gingival amount at 6 months
  The distance from the free gingival margin to the mucogingival junction was measured in millimeters with a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA).
Attached Gingival Amount | baseline attached gingival amount
  With a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA), the distance from the pocket base projection to the mucogingival junction was measured in millimeters.
Attached Gingival Amount | Change from attached gingival amount at 1 months
  With a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA), the distance from the pocket base projection to the mucogingival junction was measured in millimeters.
Attached Gingival Amount | Change from attached gingival amount at 3 months
  With a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA), the distance from the pocket base projection to the mucogingival junction was measured in millimeters.
Attached Gingival Amount | Change from attached gingival amount at 6 months
  With a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA), the distance from the pocket base projection to the mucogingival junction was measured in millimeters.
Gingival Recession Amount | baseline gingival recession amount
  The distance from the enamel-cementum border to the free gingival margin was measured in millimeters with a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA).
Gingival Recession Amount | Change from gingival recession amount at 1 months
  The distance from the enamel-cementum border to the free gingival margin was measured in millimeters with a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA).
Gingival Recession Amount | Change from gingival recession amount at 3 months
  The distance from the enamel-cementum border to the free gingival margin was measured in millimeters with a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA).
Gingival Recession Amount | Change from gingival recession amount at 6 months
  The distance from the enamel-cementum border to the free gingival margin was measured in millimeters with a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA).
Clinical Attachment Level | baseline clinical attachment level
  With a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA), the probe was inserted until a slight resistance was felt at the base of the pocket/sulcus, and the distance from the base of the pocket/sulcus to the enamel junction was measured in millimeters.
Clinical Attachment Level | Change from clinical attachment level amount at 1 months
  With a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA), the probe was inserted until a slight resistance was felt at the base of the pocket/sulcus, and the distance from the base of the pocket/sulcus to the enamel junction was measured in millimeters.
Clinical Attachment Level | Change from clinical attachment level amount at 3 months
  With a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA), the probe was inserted until a slight resistance was felt at the base of the pocket/sulcus, and the distance from the base of the pocket/sulcus to the enamel junction was measured in millimeters.
Clinical Attachment Level | Change from clinical attachment level amount at 6 months
  With a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA), the probe was inserted until a slight resistance was felt at the base of the pocket/sulcus, and the distance from the base of the pocket/sulcus to the enamel junction was measured in millimeters.
Gingival Thickness | baseline gingival thickness
  The distance from the 2 mm apical gingival margin to the hard tissue was measured in millimeters by inserting a 0.5 mm deep William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA) into the gingiva under topical anesthesia and completed to the nearest value.
Gingival Thickness | Change from gingival thickness amount at 6 months
  The distance from the 2 mm apical gingival margin to the hard tissue was measured in millimeters by inserting a 0.5 mm deep William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA) into the gingiva under topical anesthesia and completed to the nearest value.
Gingival Recession Width | baseline gingival recession width
  The mesio-distal width of the gingival recession at the level of the enamel-cementum border of the tooth was measured millimetrically with a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA).
Gingival Recession Width | Change from gingival recession width at 6 months
  The mesio-distal width of the gingival recession at the level of the enamel-cementum border of the tooth was measured millimetrically with a 0.5 mm diameter William's type periodontal probe (Nordent Manufacturing Inc, Elk Grove Village, IL, USA).
Percentage of Root Surface Coverage (%) | It was calculated using the formula at 6 months after surgical procedures.
  Baseline GRA - Postoperative 6th month GRA RCP (%) = --------------------- X 100 Baseline GRA

CONTACTS AND LOCATIONS:
Overall Officials: Kevser Sökmen, asst. prof., Principal Investigator — kevser.sokmen@alanya.edu.tr
Locations (1):
- Alanya Alaaddin Keykubat University, Faculty of Dentistry, Department of Periodontology, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
A new indication will be provided for the use of BTX-A.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: may remain open indefinitely
Access Criteria: everyone

REFERENCES:
- [Background] Goyal L, Gupta ND, Gupta N, Chawla K. Free Gingival Graft as a Single Step Procedure for Treatment of Mandibular Miller Class I and II Recession Defects. World J Plast Surg. 2019 Jan;8(1):12-17. doi: 10.29252/wjps.8.1.12.. PMID 30873357
- [Background] Dias JJ, Panwar M, Kosala M. Management of inadequate keratinized gingiva and millers class III or IV gingival recession using two-stage free gingival graft procedure. J Indian Soc Periodontol. 2020 Nov-Dec;24(6):554-559. doi: 10.4103/jisp.jisp_531_19. Epub 2020 Nov 14. PMID 33424173
- [Background] AlJasser RN, AlSarhan MA, AlOtaibi DH, AlOraini S, AlNuwaiser R, AlOtaibi A, Alduraihem H, Habib SR, Zafar MS. Comparison of Polymeric Cyanoacrylate Adhesives with Suturing in Free Gingival Graft Stability: A Split Mouth Trial. Polymers (Basel). 2021 Oct 16;13(20):3575. doi: 10.3390/polym13203575. PMID 34685335
- [Background] Freeman SR, Cohen JL. New neurotoxins on the horizon. Aesthet Surg J. 2008 May-Jun;28(3):325-30. doi: 10.1016/j.asj.2008.03.006. PMID 19083544
- [Background] Serrera-Figallo MA, Ruiz-de-Leon-Hernandez G, Torres-Lagares D, Castro-Araya A, Torres-Ferrerosa O, Hernandez-Pacheco E, Gutierrez-Perez JL. Use of Botulinum Toxin in Orofacial Clinical Practice. Toxins (Basel). 2020 Feb 11;12(2):112. doi: 10.3390/toxins12020112. PMID 32053883
- [Background] Roh TS, Jung BK, Yun I, Lew DH, Kim YS. Effect of botulinum toxin A on vasoconstriction and sympathetic neurotransmitters in a murine random pattern skin flap model. Wound Repair Regen. 2017 Jan;25(1):75-85. doi: 10.1111/wrr.12501. Epub 2017 Jan 5. PMID 27997734
- [Background] Kim TK, Oh EJ, Chung JY, Park JW, Cho BC, Chung HY. The effects of botulinum toxin A on the survival of a random cutaneous flap. J Plast Reconstr Aesthet Surg. 2009 Jul;62(7):906-13. doi: 10.1016/j.bjps.2007.12.034. Epub 2008 Apr 24. PMID 18436495
- [Background] Hull M, Parnes M. Effective Treatment of Geniospasm: Case Series and Review of the Literature. Tremor Other Hyperkinet Mov (N Y). 2020 Aug 17;10:31. doi: 10.5334/tohm.141. PMID 32874771
- [Background] Papel ID, Capone RB. Botulinum toxin A for mentalis muscle dysfunction. Arch Facial Plast Surg. 2001 Oct-Dec;3(4):268-9. doi: 10.1001/archfaci.3.4.268. PMID 11710863